CLINICAL TRIAL: NCT06766721
Title: Diagnostic Effectiveness of Ultrasound in Costochondral Joint Separation: A Prospective Study
Brief Title: Ultrasound for Diagnosing Costochondral Joint Separation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Caner İşevi, MD (Other)
Responsible Party: Sponsor-Investigator, Caner İşevi, MD, Principal Investigator, Ondokuz Mayıs University
Organization: Ondokuz Mayıs University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: B.30.2.ODM.0.20.08/517
Record Dates: First submitted 2024-12-29; First posted 2025-01-09 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2024-12

CONDITIONS: Rib Fractures; Thoracic Injuries
Keywords: Costochondral Joint Separation; Ultrasound; Blunt Thoracic Trauma; Thoracic Surgery; Computed Tomography
MeSH Terms: conditions — Rib Fractures; Thoracic Injuries | interventions — Ultrasonography

STUDY DESIGN:
Intervention Model Description: This study employs a single-group design where all participants will undergo both ultrasound (USG) and computed tomography (CT) imaging. The purpose is to evaluate the diagnostic accuracy of USG in detecting costochondral joint separation by comparing its findings with those of CT, considered the gold standard. No control or comparison groups are included in this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Diagnostic Ultrasound Evaluation (Experimental): All participants will undergo both ultrasound (USG) and computed tomography (CT) imaging as part of the diagnostic protocol. The purpose of this arm is to evaluate the diagnostic accuracy of USG in detecting costochondral joint separation. USG findings will be compared to CT results, which serve as the gold standard, to determine sensitivity, specificity, and accuracy.
  This single-arm design ensures all participants receive the same diagnostic procedures without assignment to different groups or interventions.
  Interventions: Device: Ultrasound (USG)

INTERVENTIONS:
Device: Ultrasound (USG) — The intervention involves the use of a portable ultrasound (USG) device to assess costochondral joint separation in patients with blunt thoracic trauma. The ultrasound examination will focus on detecting disruptions in the connection between the ribs and cartilage, providing a non-invasive, radiation-free diagnostic method. A 12-MHz linear transducer will be used to scan the rib area for fractures or separations. The findings will be compared to those of computed tomography (CT), considered the gold standard. This intervention is designed to evaluate the accuracy, sensitivity, and specificity of ultrasound as a diagnostic tool in this context.

SUMMARY:
This study aims to evaluate the diagnostic effectiveness of ultrasound in detecting costochondral joint separation in patients with blunt thoracic trauma. By comparing ultrasound findings to computed tomography (CT) results, the study seeks to determine the sensitivity, specificity, and overall accuracy of ultrasound as a diagnostic tool. The results will help improve the diagnosis and management of costochondral injuries while minimizing radiation exposure. The study is a prospective, interventional trial conducted at Ondokuz Mayıs University Faculty of Medicine.

DETAILED DESCRIPTION:
This study investigates the diagnostic effectiveness of ultrasound (USG) in identifying costochondral joint separation in patients presenting with blunt thoracic trauma. The study aims to assess USG's sensitivity, specificity, and accuracy compared to computed tomography (CT), which is considered the gold standard.

Costochondral separation, a condition where the connection between the rib and its cartilage is disrupted, is often challenging to diagnose with traditional imaging techniques. Ultrasound offers a non-invasive, portable, and radiation-free alternative, potentially allowing for rapid diagnosis and improved patient outcomes.

Participants will undergo both USG and CT imaging as part of the diagnostic protocol. The primary outcome measure will be the diagnostic accuracy of USG in detecting costochondral joint separation. Secondary outcomes include time to diagnosis, patient comfort, and correlation of ultrasound findings with clinical presentations.

The study will be conducted prospectively at Ondokuz Mayıs University Faculty of Medicine from March 2025 to March 2027, involving a sample size of 51 patients based on power analysis. Data collected will include demographic information, trauma specifics, imaging findings, and clinical outcomes.

The results are expected to contribute significantly to the field of thoracic trauma care by demonstrating the utility of ultrasound in settings where quick and accurate diagnosis is critical.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 80 years
* Patients with blunt thoracic trauma
* Patients suspected of having costochondral joint separation
* Patients who provide consent for ultrasound and CT imaging

Exclusion Criteria:

* Patients under 18 or over 80 years of age
* Patients with penetrating thoracic trauma
* Patients with subcutaneous emphysema that prevents ultrasound evaluation
* Patients allergic to ultrasound gel
* Pregnant patients (as CT imaging is contraindicated)
* Patients unable to undergo CT imaging
* Patients who refuse to participate in the study
* Obese patients (body mass index >30), as ultrasound evaluation may be challenging

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Accurate Ultrasound Diagnosis Compared to CT | Within the first 24 hours of patient admission.
  The diagnostic accuracy (sensitivity, specificity, and overall accuracy) of ultrasound (USG) in detecting costochondral joint separation, using computed tomography (CT) as the reference standard.

CONTACTS AND LOCATIONS:
Locations (1):
- Ondokuz Mayıs University, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Stengel D, Leisterer J, Ferrada P, Ekkernkamp A, Mutze S, Hoenning A. Point-of-care ultrasonography for diagnosing thoracoabdominal injuries in patients with blunt trauma. Cochrane Database Syst Rev. 2018 Dec 12;12(12):CD012669. doi: 10.1002/14651858.CD012669.pub2. PMID 30548249
- [Background] Wilkerson RG, Stone MB. Sensitivity of bedside ultrasound and supine anteroposterior chest radiographs for the identification of pneumothorax after blunt trauma. Acad Emerg Med. 2010 Jan;17(1):11-7. doi: 10.1111/j.1553-2712.2009.00628.x. PMID 20078434